CLINICAL TRIAL: NCT05193565
Title: Multi-center, Open-label, Randomized Controlled Phase 4 Study to Compare the Efficacy and Safety After Conversion to RaparoBell® or My-Rept® in Kidney Transplant Patients Undergoing Maintenance Therapy With CNI Plus MPA.[CORAL Study]
Brief Title: Study to Compare the Efficacy and Safety After Conversion to RaparoBell® or My-Rept® in Kidney Transplant Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B110_02KT2103
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2021-12

CONDITIONS: Kidney Transplantation
Keywords: Kidney Transplantation; Sirolimus
MeSH Terms: interventions — Sirolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RaparoBell Tablet (Experimental): RaparoBell Tablet
  Interventions: Drug: Sirolimus
- Mycophenolate Mofetil Tablet/Capsule (Active Comparator): Myrept Tablet/Capsule
  Interventions: Drug: Mycophenolate mofetil

INTERVENTIONS:
Drug: Sirolimus — Orally, once-daily in the morning - Check the blood concentration of Sirolimus at each visit and adjust the dose to achieve the blood concentration maintaining at 3~8ng/mL
  Other Names: RaparoBell® Tab.
  Arms: RaparoBell Tablet
Drug: Mycophenolate mofetil — Up to 1g BID(total 2g daily), PO
  Other Names: Myrept® Cap./Tab.
  Arms: Mycophenolate Mofetil Tablet/Capsule

SUMMARY:
The purpose of this study is to evaluate the efficacy and Safety after conversion to RaparoBell® or Myrept® in patients who in renal transplant patients undergoing maintenance therapy with Mycophenolic acid.

DETAILED DESCRIPTION:
This study is a multi-center, Randomized, Open-label and phase IV clinical trial that evaluates the efficacy and safety after conversion to RaparoBell® or Myrept® administration for 24 weeks in renal transplant patients undergoing maintenance therapy with Mycophenolic acid.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who at least 1 year and less than 10 years after kidney transplantation
2. Over 20 years old
3. Patients on immunosuppressive maintenance therapy using combination of Calcineurin Inhibitor and Mycophenolic acid after kidney transplantation

Exclusion Criteria:

1. Patients who have transplanted organs other than kidney
2. At the time of Screening

   * Treatment with active liver disease or Liver function test(T-bilirubin, AST, ALT)is over 3 times than upper normal limit
   * WBC< 2,500/mm^3, or platelet < 75,000/mm^3, or ANC < 1,300/ mm^3
   * Protein/Creatinine ratio≥1.0(mg/mg)
3. Patents who had a record of taking mTOR inhibitor before 3 months
4. In investigator's judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2021-11-19 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of composite efficacy failure | Until 24 weeks
  Composite efficacy failure include biopsy-confirmed acute rejection, graft loss, death, or follow-up failure

SECONDARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection(TCMR, AMR) | Until 24 weeks
  The frequency and Incidence
Pathologic Results, Occurrence, Treatment Methods, and Results of Acute Rejection Confirmed by Biopsy | Until 24 weeks
  By Banff classification categories
Survival rate of transplanted organ | Until 24 weeks
  Kaplan-Meier
Survival rate of Patients | Until 24 weeks
  Kaplan-Meier
Serum-Cr, eGFR | Until 24 weeks
  eGFR using MDRD
Incidence of BKV, CMV infection | Until 24 weeks
  The frequency and Incidence

CONTACTS AND LOCATIONS:
Overall Officials: Chul Woo Yang, Ph.D, Study Chair — The Catholic University of Korea
Locations (1):
- The Catholic University of Korea, Seoul, St.Mary's Hospital, Seoul, South Korea